CLINICAL TRIAL: NCT01730833
Title: Phase II Prospective Open Label Study of Pertuzumab, Trastuzumab, and Nab-Paclitaxel in Patients With HER-2 Positive Advanced Breast Cancer
Brief Title: Pertuzumab, Trastuzumab, and Paclitaxel Albumin-Stabilized Nanoparticle Formulation in Treating Patients With HER2-Positive Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12147; NCI-2012-02371 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA166020 (NIH); AACR Grant 12-60-26-WANG (Other Grant/Funding Number: Breast Cancer Research Foundation)
Record Dates: First submitted 2012-11-16; First posted 2012-11-21 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: HER2-positive Breast Cancer; Recurrent Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer; Breast Adenocarcinoma; Inflammatory Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — pertuzumab; 2C4 antibody; Trastuzumab; Taxes; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pertuzumab, trastuzumab, nab-paclitaxel) (Experimental): Patients receive pertuzumab IV over 30-60 minutes on day 1, trastuzumab IV over 30-90 minutes and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: pertuzumab; Biological: trastuzumab; Drug: paclitaxel albumin-stabilized nanoparticle formulation; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: pertuzumab — Given IV
  Other Names: 2C4 antibody; monoclonal antibody 2C4; Perjeta; rhuMAb-2C4
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: paclitaxel albumin-stabilized nanoparticle formulation — Given IV
  Other Names: ABI-007; nab paclitaxel; nab-paclitaxel; nanoparticle albumin-bound paclitaxel
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial studies how well pertuzumab, trastuzumab, and paclitaxel albumin-stabilized nanoparticle formulation work in treating patients with human epidermal growth factor receptor (HER) 2-positive stage II-IV breast cancer. Monoclonal antibodies, such as pertuzumab and trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation, work in different ways to kill tumor cells or stop them from growing. Giving pertuzumab and trastuzumab together with paclitaxel albumin-stabilized nanoparticle formulation may be a better way to block tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine efficacy of administration of pertuzumab in combination with trastuzumab with nab-paclitaxel (paclitaxel albumin-stabilized nanoparticle formulation) in subjects with stage IV human epidermal growth factor receptor (HER)-2 overexpressing metastatic breast cancer (MBC) as measured by progression free survival (PFS).

II. To determine the efficacy as neoadjuvant treatment of the regimen in HER2+ locally advanced breast cancer (LABC) as defined by pathologic complete response (pCR).

SECONDARY OBJECTIVES:

I. To evaluate the safety of pertuzumab when added to trastuzumab and nab-paclitaxel in HER-2 overexpressing MBC and LABC cancer as assessed by the frequency and severity of adverse events (AEs), abnormal findings on physical examination, laboratory tests, and vital signs.

II. To evaluate the objective response rate (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) and duration of response in MBC.

III. To evaluate the efficacy of the regimen by assessing tumor response including assessment of residual cancer burden (RCB) scores in LABC.

IV. To assess the progression free survival (MBC), relapse-free survival (LABC) and overall survival in all patients.

V. To perform exploratory circulatory gene, micro-ribonucleic acid (RNA), and exosome profiling as well as protein and glycomic profiling.

VI. To assess the feasibility of molecular profiling in both primary and metastatic tumor samples.

VII. To assess numerical and qualitative aspects of circulating tumor cells and circulating tumor-derived deoxyribonucleic acid (DNA).

OUTLINE: Patients receive pertuzumab intravenously (IV) over 30-60 minutes on day 1, trastuzumab IV over 30-90 minutes and paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity (patients with MBC) or for 6 courses in the absence of disease progression or unacceptable toxicity (patients with LABC).

After completion of study treatment, patients are followed up every 3 months for 4 years and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with metastatic cytologically or histologically confirmed adenocarcinoma of the breast with HER2 over-expression or with newly diagnosed locally advanced (including inflammatory) breast cancer (LABC) with stage II-III disease; patients with metastatic (stage IV) disease (MBC) must have measurable lesions
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* Tumor positive or negative for expression of hormone receptors (< 1% or > 1%) and overexpressing HER2 by immunohistochemistry (IHC) (3+), or, HER2-amplified by fluorescence in situ hybridization (FISH) or by alternative gene testing
* For patients with LABC, no prior therapy is allowed
* For patients with MBC, prior adjuvant chemotherapy and trastuzumab more than or equal to 12 months prior to enrollment are allowed
* No prior chemotherapy or trastuzumab for treatment of metastatic breast cancer
* Left ventricular ejection fraction (LVEF) >= 50% (determined by echocardiogram or multigated acquisition scan) within 42 days of treatment
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Hemoglobin >= 9 g/dl
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< 1.3 mg/dl (institutional upper limit of normal)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance > 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (using Cockcroft-Gault formula)
* All radiology studies (study requiring staging) must be performed within 35 days prior to the start of therapy
* No serious medical conditions such as myocardial infarction within 6 months prior to entry, congestive heart failure, unstable ventricular arrhythmia, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled psychotic disorders, serious infections, active peptic ulcer disease, psychiatric illness, or any other medical conditions that might be aggravated by treatment or limit compliance
* Currently, no active second malignancy other than non-melanoma skin cancer; note: patients are not considered to have a "current active" malignancy if they have completed anti-cancer therapy and are considered by their physicians to have a less than 30% chance of relapse
* All patients must have the ability to understand and the willingness to sign an informed consent
* Negative serum or urine beta-human chorionic gonadotropin (hCG) pregnancy test at screening for patients of child-bearing potential
* No prior therapies (except for anti-estrogen therapy) are allowed for the treatment of the newly diagnosed metastatic breast cancer; patients are allowed to have had prior chemotherapy for breast cancer in the adjuvant setting for at least 12 months prior to enrollment into this study; patients with a prior diagnosis of malignancy treated >= 5 years ago are eligible, provided that they have not received prior nab-paclitaxel as part of their prior treatment regimen, and that they meet all eligibility criteria

Exclusion Criteria:

* Known active hepatitis B or C
* Known active human immunodeficiency virus (HIV)
* Prior breast cancer or other invasive malignancy treated within 5 years
* Pregnancy
* Neuropathy > grade 1
* Any other intercurrent medical/psychological problem deemed exclusionary by the treating physician or investigators/principal investigator (PI)
* Cumulative dose of doxorubicin or equivalent of > 360 mg/m^2 during prior adjuvant therapy
* LVEF < 50% during previous trastuzumab therapy
* Central nervous system metastases
* Another malignancy excluding basal cell skin cancer
* Pregnant women
* Subjects will be excluded who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-07-17 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2026-05-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Mortimer, MD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope- South Pasadena Cancer Center, South Pasadena, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients: Pertuzumab administered as 840 mg IV during cycle 1 followed by 420 mg IV once every three weeks starting cycle 2.
  Trastuzumab loading dose of 4mg/kg IV for week one followed by 2mg/kg IV weekly.
  Nab-paclitaxel 100 mg/m2 IV weekly.
  Treatment is scheduled to continue until:
  Disease progression Unmanageable toxicity Primary physician or patient request to discontinue therapy Study termination by the sponsors
- Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients: Pertuzumab administered as 840 mg IV during cycle 1 followed by 420 mg IV once every three weeks starting cycle 2.
  Trastuzumab loading dose of 4mg/kg IV for week one followed by 2mg/kg IV weekly.
  Nab-paclitaxel 100 mg/m2 IV weekly.
  Treatment is scheduled to continue until:
  A planned 6 cycles Unmanageable toxicity Primary physician or patient request to discontinue therapy Study termination by the sponsors
Period: Overall Study
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients
Started | 18 | 45
Completed | 18 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients | Total
Number analyzed (Participants) | 18 | 45 | 63
Age, Continuous [Median (Full Range); unit: years] | 49 [31 to 65] | 56 [31 to 78] | 54 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 45 | 63
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 1 | 2
  Asian | 2 | 7 | 9
  Hispanic | 10 | 19 | 29
  Non-Hispanic White | 5 | 17 | 22
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 18 | 45 | 63

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (MBC Cohort)
Description: Estimated using the product-limit method of Kaplan and Meier. From time of initial treatment until disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: assessed up to 5 years
Population: PFS was not performed on the LABC cohort (neoadjuvant patients). A more relevant analysis, Disease-free survival is present elsewhere in these results.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients
Number analyzed (Participants) | 18 | 0
Months | 22.4 [7.1 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. |

2. Primary Outcome: Five Year Disease-free Survival (LABC Cohort)
Description: Estimated using the method of Kaplan-Meier. Disease-free survival is defined as the time from Initial treatment to recurrence of tumor or death
Time Frame: assessed up to 5 years
Population: Analysis population included LABC participants who achieved pathologic response (pCR). More appropriate PFS analysis for MBC cohort is presented elsewhere in these results.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients
Number analyzed (Participants) | 0 | 29
percentage of participants |  | 96.3 [76.5 to 99.5]

3. Secondary Outcome: Overall Response (MBC Cohort)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 5 years
Population: Overall response is not appropriate in the neoadjuvant or LABC cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients
Number analyzed (Participants) | 18 | 0
Participants | 13 |

4. Secondary Outcome: Five Year Overall Survival
Description: Estimated by the Kaplan-Meier method. From the initial date of treatment to date of death from any cause.
Time Frame: Assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients
Number analyzed (Participants) | 18 | 45
percentage of participants | 54.5 [8.6 to 86.1] | 94.1 [77.6 to 98.5]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time of initial treatment until 30 days post discontinuation of treatment, up to 5 years.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients
All-Cause Mortality (participants affected / at risk) | 8/18 | 2/45
Serious Adverse Events (participants affected / at risk) | 3/18 | 4/45
Other Adverse Events (participants affected / at risk) | 18/18 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients (N=18) | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients (N=45)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Oth (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (6) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort1: Stage IV HER-2 Overexpressing Metastatic Breast Cancer (MBC) Patients (N=18) | Cohort 2: HER2+ Locally Advanced Breast Cancer (LABC) Patients (N=45)
Anemia (Blood and lymphatic system disorders) | 16 (162) | 40 (172)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (4)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 2 (6) | 2 (7)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 6 (21) | 7 (22)
Tricuspid valve disease (Cardiac disorders) | 1 (2) | 0 (0)
Ear and labyrinth disorders - Other, spe (Ear and labyrinth disorders) | 0 (0) | 1 (4)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (3)
Vestibular disorder (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 5 (12) | 2 (2)
Dry eye (Eye disorders) | 2 (3) | 3 (7)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 4 (6)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (2) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 7 (11)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 8 (12) | 16 (34)
Diarrhea (Gastrointestinal disorders) | 10 (29) | 31 (86)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (5)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (20) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (6) | 5 (15)
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 2 (3) | 6 (8)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (23) | 8 (22)
Mucositis oral (Gastrointestinal disorders) | 5 (14) | 8 (14)
Nausea (Gastrointestinal disorders) | 8 (24) | 28 (68)
Oral dysesthesia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (2) | 3 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1) | 2 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (8) | 10 (12)
Chills (General disorders) | 1 (2) | 7 (7)
Edema face (General disorders) | 1 (2) | 1 (3)
Edema limbs (General disorders) | 10 (62) | 17 (39)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 16 (120) | 43 (183)
Fever (General disorders) | 2 (2) | 5 (7)
Flu like symptoms (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 2 (3) | 0 (0)
General disorders and administration sit (General disorders) | 0 (0) | 1 (3)
Infusion related reaction (General disorders) | 5 (6) | 7 (9)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 2 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 4 (10) | 6 (11)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Breast infection (Infections and infestations) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (2) | 1 (2)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 2 (8) | 6 (13)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 5 (29) | 5 (7)
Rash pustular (Infections and infestations) | 1 (3) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (4)
Skin infection (Infections and infestations) | 1 (1) | 2 (5)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (12) | 7 (12)
Urinary tract infection (Infections and infestations) | 2 (2) | 5 (7)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (5) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (4) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 11 (27) | 22 (79)
Alkaline phosphatase increased (Investigations) | 3 (8) | 9 (24)
Aspartate aminotransferase increased (Investigations) | 10 (44) | 16 (62)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 0 (0) | 2 (5)
Creatinine increased (Investigations) | 0 (0) | 2 (7)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 4 (5)
Lymphocyte count increased (Investigations) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 8 (29) | 13 (26)
Platelet count decreased (Investigations) | 3 (4) | 2 (7)
Serum amylase increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 2 (4) | 2 (3)
Weight loss (Investigations) | 1 (1) | 3 (10)
White blood cell decreased (Investigations) | 14 (108) | 27 (80)
Anorexia (Metabolism and nutrition disorders) | 5 (10) | 7 (17)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (9) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 4 (6) | 7 (14)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (23) | 7 (13)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (29) | 8 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (11) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 5 (15) | 12 (26)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (13) | 16 (33)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3) | 8 (16)
Metabolism and nutrition disorders - Oth (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 5 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (9) | 3 (9)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (20) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (12) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 8 (13)
Neoplasms benign, malignant and unspecif (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (13) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (7) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (7) | 13 (31)
Headache (Nervous system disorders) | 6 (18) | 7 (8)
Nervous system disorders - Other, specif (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 2 (2) | 4 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 15 (104) | 36 (150)
Spasticity (Nervous system disorders) | 2 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (17) | 8 (17)
Depression (Psychiatric disorders) | 3 (8) | 4 (11)
Insomnia (Psychiatric disorders) | 6 (16) | 8 (22)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 2 (3) | 5 (10)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 2 (5)
Menorrhagia (Reproductive system and breast disorders) | 2 (5) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (18) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (16) | 10 (18)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (12) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 9 (17)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 6 (8)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (73) | 16 (42)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (8) | 10 (22)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 5 (37) | 15 (38)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (16) | 3 (8)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (5) | 3 (5)
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (9) | 10 (19)
Rash acneiform (Skin and subcutaneous tissue disorders) | 9 (46) | 24 (78)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (9) | 11 (24)
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 8 (30) | 13 (30)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 8 (43) | 12 (34)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hot flashes (Vascular disorders) | 2 (3) | 6 (21)
Hypertension (Vascular disorders) | 14 (122) | 29 (148)
Hypotension (Vascular disorders) | 1 (2) | 4 (4)
Lymphedema (Vascular disorders) | 3 (7) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (4) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/33/NCT01730833/Prot_SAP_000.pdf